CLINICAL TRIAL: NCT05098808
Title: Classification of Dysphagia Patients at Risk of Aspiration Pneumonia Using Machine Learning Algorithms Incorporating Acoustic Features From Phonetic Evaluation
Brief Title: Artificial Intelligence in Diagnosing Dysphagia Patients
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sun Im, associate professor, The Catholic University of Korea
Other Study IDs: HC19EESE0060
Record Dates: First submitted 2021-10-01; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Respiration Disorders; Swallowing Disorder; Phonation Disorder; Stroke; Aspiration Pneumonia; Aspiration; Liquids
MeSH Terms: conditions — Respiration Disorders; Deglutition Disorders; Dysphonia; Stroke; Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysphagia mild: Able to start oral feeding after assessment
  Interventions: Other: Acoustic features (from signals obtained during phonation)
- Dysphagia severe: Non oral feeding and high risk of aspiration
  Interventions: Other: Acoustic features (from signals obtained during phonation)

INTERVENTIONS:
Other: Acoustic features (from signals obtained during phonation) — Acoustic features will be obtained via phonation files.
  A voice recorder application provided by Apple was used, and the sampling frequency of the sound was 44,100 Hz. The digitized cough sound signals were band-pass-filtered between 20 to 16,000 Hz to use data from the whole frequency band gathered by the iPad. In each case, the smart device was positioned 20cm from the patient

SUMMARY:
In this prospective study we extracted acoustic parameters using PRAAT from patient's attempt to phonate during the clinical evaluation using a digital smart device. From these parameters we attempted (1) to define which of the PRAAT acoustic features best help to discriminate patients with dysphagia (2) to develop algorithms using sophisticated ML techniques that best classify those i) with dysphagia and those ii ) at high risk of respiratory complications due to poor cough force.

DETAILED DESCRIPTION:
This study was prospective study, and patients who visited the department of rehabilitation medicine in a single university-affiliated tertiary hospital with dysphagic symptoms from September 2019 to March 2021 were included.Voice recording was performed at the enrollment with blinded assessment, where the participants first visited the rehabilitation department with chief complaints of dysphagia. The cough sounds were recorded with an iPad (Apple, Cupertino, CA, USA) through an embedded microphone.

From the acoustic files we extracted fourteen voice parameters that include the average value and standard deviation of the fundamental frequency (f0), harmonic-to-noise ratio (HNR), the jitter that refers to frequency instability, and the shimmer that represents the amplitude instability of the sound signal.

Machine learning algorithms and sophisticated deep neural network analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria

1. Suspected swallowing disorder who were referred for swallowing assessment
2. Dysphagia attributable to brain lesion including stroke

Exclusion Criteria:

1. Participants who were unable to perform phonation
2. Participants who had no VFSS or standardized swallowing assessment results
3. Participants with no spirometric measurements

Ages: 19 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: First ever stroke patients referred for swallowing disorders
Sampling Method: Non-Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Functional Oral Intake Scale | during the intervention
  Dysphagia severity as measured by the the Functional Oral Intake Scale obtained from standardized swallowing tests
Cough strength | during the intervention
  Spirometry values : cough strength as measured by the spirometric values during voluntary cough

CONTACTS AND LOCATIONS:
Overall Officials: Sun Im, MD PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Department of Rehabilitation Medicine Bucheon St Mary's Hospital, Catholic University of Korea, College of Medicine, Bucheon-si, Kyounggido, South Korea

IPD SHARING:
Plan to Share IPD: No
Data would be accessible only upon formal request to the formal PI